CLINICAL TRIAL: NCT07353216
Title: Exploring the Efficacy and Safety of Ofatumumab in Patients With Relapsing Multiple Sclerosis (RMS) and Its Impact on Serum Neurofilament Light Chain (sNfL) Levels：A Multicenter, Open-Label, Observational Real-World Study
Brief Title: Exploring the Efficacy and Safety of Ofatumumab in Patients With Relapsing Multiple Sclerosis (RMS) and Its Impact on Serum Neurofilament Light Chain (sNfL) Levels
Status: Recruiting | Type: Observational
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Shenzhen Second People's Hospita (Unknown); Shenzhen People's Hospital (Other)
Responsible Party: Principal Investigator, Wei Qiu, Chief Physician, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: 2023-305-01
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: NfL, Multiple sclerosis, treatment
MeSH Terms: conditions — Multiple Sclerosis | interventions — ofatumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ofatumumab — Ofatumumab 20mg

SUMMARY:
Multiple sclerosis (MS) is an immune-mediated disease characterized primarily by inflammatory demyelinating lesions in the central nervous system (CNS), with the white matter being predominantly affected. Its etiology remains unclear and may be associated with various factors such as genetics, environment, and viral infections . Pathologically, MS presents as multiple demyelinating lesions in the CNS, which may be accompanied by damage to nerve cells and their axons. Lesions on MRI show characteristic distributions, morphologies, and signal intensities . MS typically onset in young adults and is more common in women. Frequent symptoms include visual decline, diplopia, limb sensory disturbances, limb motor impairment, ataxia, and bladder or rectal dysfunction . As MS can lead to varying degrees of neurological deficits, and repeated relapses result in disability progression, it impacts patients' normal lives and work, posing a significant burden on individuals, families, and society. Considerable progress has been made in MS treatment in recent years, with agents such as teriflunomide, fingolimod, siponimod, and dimethyl fumarate having been approved for marketing in China.

In the two concurrently conducted active-comparator trials, ASCLEPIOS I and II, involving patients with relapsing multiple sclerosis, the annualized relapse rate was significantly lower in the ofatumumab group compared to the teriflunomide group. Ofatumumab was also superior to teriflunomide in suppressing MRI lesion activity . Although the aforementioned studies have confirmed the clinical efficacy of ofatumumab in treating MS, data from Chinese populations are lacking. Its clinical effectiveness, safety, and optimal treatment timing require further support from real-world evidence.

Exploring more indicators to predict MS disease activity and progression is crucial for identifying high-risk patients, assessing prognosis, and evaluating treatment response. Neurofilament light chain (NfL) is a specific biomarker for neuroaxonal damage, released into the cerebrospinal fluid (CSF) and serum after axonal injury . Serum and CSF NfL concentrations are highly correlated. Numerous studies in recent years have shown that high sNfL levels are associated with active T2 lesions and relapses, as well as brain volume loss. sNfL can not only monitor disease activity and treatment response at the group level in MS patients but also predict disease course, making it a valuable biomarker for predicting MS relapses and disability progression. It helps identify patients at higher risk of future disease activity and assists in clinical decision-making. Previous data from ASCLEPIOS I and II demonstrated that ofatumumab significantly reduced sNfL concentrations at the first assessment (Month 3) and at all subsequent visits in patients with RMS . However, existing studies have not included data from Chinese populations. This study aims to address this data gap for this specific population.

ELIGIBILITY:
Inclusion Criteria:Signed and dated informed consent must be obtained before participation in the study.

Any gender, aged at least 18 years at the time of study enrollment (signing the informed consent form).

Patients with RMS meeting the 2017 Revised McDonald Criteria. EDSS score between 0 and 7. Regular follow-up with MRI monitoring. Willingness to provide blood samples. Willingness to undergo clinical assessments (including scales and physical examinations).

-

Exclusion Criteria:Decision by the subject/legal guardian . Pregnancy. Diagnosis of Progressive Multifocal Leukoencephalopathy (PML). Hypersensitivity reaction to the investigational drug. Protocol violation that poses a significant safety risk to the subject. Occurrence of certain adverse events, such as malignancy, hepatic failure, or severe chronic infections (e.g., active hepatitis B, HIV).

Any laboratory abnormality that, considering the subject's overall condition, is deemed to prevent the subject's continued participation in the study.

Any condition that may pose a safety risk due to participation in the study. Non-compliance with the administration of the investigational drug or study procedures

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: gender unrestricted, aged at least 18 years, diagnosed with Relapsing Multiple Sclerosis (RMS)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Ofatumumab treatment reduces sNfL levels in patients with Relapsing Multiple Sclerosis | Evaluation timing includes from the baseline to 12 and 24 months after starting Ofatumumab treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No